CLINICAL TRIAL: NCT03794479
Title: Changes in Intestinal Microbiota and Acquisition of Antimicrobial Resistance in Hong Kong Residents After Travel
Brief Title: Intestinal Microbiota and Antimicrobial Resistance in Hong Kong Residents After Travel
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: travellers_version 2_20180724
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Antimicrobial Resistance
Keywords: Intestinal microbiota; Antimicrobial resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Travellers: Adults planning for travel

SUMMARY:
International travel is well reported to be associated with acquisition of multidrug-resistant organisms, however, the impact of colonization of these multidrug-resistant organisms is currently uncertain. As colonization of multidrug-resistant organisms had been demonstrated to be associated with distinct intestinal microbiota composition and travellers constitute a generally healthy population with minimal antibiotics exposure; by evaluating serial stool samples before and after travel, the investigators can delineate a potential causal relationship between host intestinal microbiota and subsequent risk of acquisition of multidrug-resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Chinese ethnicity
* Planning to visit any places outside of Hong Kong within the next three months
* Able to provide informed consent

Exclusion Criteria:

* Use of antibiotics within 4 weeks prior to the time of recruitment (Except for antimalarial prophylaxis)
* Hospitalization within 3 months
* Underlying gastrointestinal diseases, including gastrointestinal malignancy, inflammatory bowel disease, resection of small or large bowel
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults planning for travel
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients acquiring intestinal colonization of ESBL-producing Enterobacteriaceae | 1 year
  Intestinal colonization of ESBL-producing Enterobacteriaceae is defined as the presence of ESBL in Enterobacteriaceae identified in the post-travel stool samples, in patients without these organisms detected in their stool samples before travel.

SECONDARY OUTCOMES:
Proportion of patients acquiring intestinal colonization of carbapenem-resistant Enterobacteriaceae | 1 year
  Intestinal colonization of carbapenem-resistant Enterobacteriaceae is defined as the presence of carbapenem-resistant Enterobacteriaceae identified in the stool samples, in patients without these organisms detected in their stool samples before travel.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided